CLINICAL TRIAL: NCT06788743
Title: Impact of Sevoflurane Versus Propofol on Postoperative Delirium in Elderly Diabetic Patients Undergoing Non-Cardiac Surgery: a Multicenter, Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCT06788743
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Delirium (POD); Diabetes
MeSH Terms: conditions — Emergence Delirium; Diabetes Mellitus | interventions — Anesthesia; Propofol; Remifentanil; Sevoflurane

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TIVA (Experimental): Participants assigned to the TIVA group will receive propofol combined with remifentanil for anesthesia maintenance during the surgery
  Interventions: Drug: TIVA ( anesthesia with propofol and remifentanil)
- VA (Experimental): Participants assigned to the VA group will receive sevoflurane combined with remifentanil for anesthesia maintenance during the surgery.
  Interventions: Drug: VA（anesthesia with sevoflurane and remifentanil）

INTERVENTIONS:
Drug: TIVA ( anesthesia with propofol and remifentanil) — Participants assigned to the TIVA group will receive propofol combined with remifentanil for anesthesia maintenance during the surgery
  Arms: TIVA
Drug: VA（anesthesia with sevoflurane and remifentanil） — Participants assigned to the VA group will receive sevoflurane combined with remifentanil for anesthesia maintenance during the surgery.
  Arms: VA

SUMMARY:
The present study is a multicenter， randomized controlled clinical trial, which plans to enroll 450 diabetic patients aged more than 60 years. The participants will be randomly assigned in a 1:1 ratio and will receive either propofol or sevoflurane for intraoperative anesthesia maintenance to evaluate the impact of these two anesthetic drugs on postoperative delirium. The aim of our study is to explore whether the use of propofol for anesthesia maintenance in elderly diabetic patients undergoing elective non-cardiac major surgery can reduce the incidence of postoperative delirium. This study will provide new perspectives for improving perioperative management in elderly diabetic patients and optimizing anesthesia management strategies to reduce the risk of postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years
* Elective surgery (with an expected duration of 2 hours or more)
* ASA grade Ⅰ-Ⅲ
* Voluntary participation and informed consent obtained
* Diabetes mellitus

Exclusion Criteria:

* Known neurological or psychiatric diseases (Parkinson's disease, depression, schizophrenia), or cognitive impairment (dementia)
* Severe visual or auditory impairments, language barriers, or patients who cannot cooperate
* Long-term use of sedatives, antipsychotic drugs, or long-term alcohol abuse
* Neurosurgical patients
* Patients who are expected to require hepatic portal blockage during surgery
* Patients who are expected to be transferred to ICU after surgery
* Patients with a known allergy to the drugs used in this study or those suspected of having propofol infusion syndrome

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of delirium | within the first 7 postoperative days
  Postoperative delirium will be assessed daily at 8:00 AM and 6:00 PM from postoperative days 1 to 7, or until discharge, using the 3D-CAM scale.

SECONDARY OUTCOMES:
The severity of POD | within the first 7 postoperative days
  The severity of postoperative delirium will be evaluated with the 4-item CAM-S scale (total score: 7 points, where 0 points indicates no delirium; 1 point indicates mild delirium; 2 points indicates moderate delirium; 3-7 points indicate severe delirium).
The duration of POD | within the first 7 postoperative days
  The total number of days with positive results.
The length of hospital stay | the first 7 postoperative days
Blood glucose levels | before anesthesia induction (T0), 1 h and 2 h after incision (T1, T2), at skin closure (T3), before PACU discharge (T4), and on post-operative days 1 and 2 (T5, T6)
  During the surgery, bedside capillary blood glucose levels will be measured using a portable blood glucose meter (capillary blood).

OTHER OUTCOMES:
Serum insulin levels | at 1 h and 2 h post-operatively (T1, T2)
Serum inflammatory factor (IL-6) levels | post-operative days 1 and 2 (T5, T6)
Serum neurodegenerative factor (S-100β protein) levels | post-operative days 1 and 2 (T5, T6)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Air Force Medical University, Xi’an, Shanxi, China